CLINICAL TRIAL: NCT04719455
Title: Adherence Improving Self-Management Strategy (AIMS) in Breast Cancer Patients Using Adjuvant Endocrine Treatment (AET): a Randomised Controlled Trial
Brief Title: Adherence Improving Self-Management Strategy (AIMS) in Breast Cancer Patients Using Adjuvant Endocrine Treatment (AET)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL74126.091.20
Record Dates: First submitted 2020-12-28; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention treatment experienced patients (Experimental): AIMS
  Interventions: Behavioral: Adherence Improving self-Management Strategy
- Intervention starting patients (Experimental): AIMS
  Interventions: Behavioral: Adherence Improving self-Management Strategy
- Control group treatment experienced patients (Other): Regular care
  Interventions: Other: Regular care
- Control group starting patients (Other): Regular care
  Interventions: Other: Regular care

INTERVENTIONS:
Behavioral: Adherence Improving self-Management Strategy — An in-person delivered intervention imbedded in regular follow-up care during 9-months. Patients will receive an electronic monitoring System to track medication intake and a pedometer to count daily amount of steps. During the baseline visit, the health care professional (HCP) will use pre-tested materials for informing and motivating patients; and collaboratively set goals and plans for medication adherence and physical activity. During regular follow-up consultations with the HCP, personalized visual reports of medication intake and amount of steps will be evaluated to enhance patients awareness of their (non-)adherence and (in)activity and identify any problems and solutions to reduce undesired behaviour. The control group will receive usual treatment only.
  Arms: Intervention starting patients; Intervention treatment experienced patients
Other: Regular care — Treatment as usual (appointments with nurse/nurse practioner with regular content)
  Arms: Control group starting patients; Control group treatment experienced patients

SUMMARY:
Background of the study:

Breast cancer is the most prevalent cancer in Dutch women. Adjuvant endocrine therapy (AET) substantially improves chances for survival after primary breast cancer. In practice, many women experience difficulties to adhere to treatment: besides missing single or multiple doses of medication, up to 50% of patients stop treatment prematurely due to decreased treatment motivation over time and burden of side effects. Together with patients and health care professionals, we adapted a cost-effective behavior change intervention (AIMS) for women using adjuvant endocrine therapy after breast cancer to an add-on module in regular follow up care.

Objective of the study:

The primary aim of this study is to pilot test the feasibility of the AIMS-AET intervention versus usual treatment on medication adherence in breast cancer survivors on adjuvant endocrine therapy. Intervention effects on psychosocial determinants and user experiences will be evaluated. The feasibility of testing the AIMS-AET intervention in a bigger RCT will be assessed. The secondary objective is to assess (preliminary) intervention effects on adherence, physical activity and on quality of life.

Study design:

A pilot randomised controlled trial comparing AIMS AET to usual care with an extensive mixed-methods process evaluation.

Study population:

Female outpatients of 2 Dutch hospitals with a prescription for adjuvant endocrine therapy after primary breast cancer. Intervention (if applicable):

An in-person delivered intervention imbedded in regular follow-up care during 9-months. Patients will receive an electronic monitoring System to track medication intake and a pedometer to count daily amount of steps. During the baseline visit, the health care professional (HCP) will use pre-tested materials for informing and motivating patients; and collaboratively set goals and plans for medication adherence and physical activity. During regular follow-up consultations with the HCP, personalized visual reports of medication intake and amount of steps will be evaluated to enhance patients awareness of their (non-)adherence and (in)activity and identify any problems and solutions to reduce undesired behaviour. The control group will receive usual treatment only.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* estrogen receptor positive
* diagnosis of primary breast cancer and active prescription of tamoxifen or aromatase inhibitors
* Not being treated with adjuvant endocrine therapy earlier (except voor neo-adjuvant endocrine therapy)
* started with adjuvant endocrine therapy in the last 4 weeks OR already taking adjuvant endocrine therapy (>=3 months; remaining treatment duration minimal 2 years)
* age minimal 18 years
* Able to come to the outpatient ward of the hospital for appointments with the nurse or nurse practitioner
* Able to understand Dutch or having the possibility to bring someone who translates

Exclusion Criteria:

* Not able to sign informed consent.
* Currently being treated with neo adjuvant endocrine therapy
* distant metastases proven by a positron emission tomograph (PET) scan with fluordeoxyglucose (FDG) scan
* Other invasive malignancy, except for a malignancy being treated without chemotherapy more than 5 years ago and without evidence for recurrence. Patients with basal cell or plaveisel cell skin cancer are eligible for the study.
* Participation in another interventional study for adherence or physical activity
* Treatment with ovarian suppression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-12-13 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention effects on psychosocial determinants (beliefs, motivation, social norm) | change from baseline at 12 months
  degree of agreement with statements about beliefs and motivation towards treatment and social norm assessed with a self-developed questionnaire
Intervention effects on self-efficacy | change from baseline at 12 months
  degree of agreement with statements about self-efficacy regarding treatment measured with the Self Efficacy of Appropriate Medication use Scale (SEAMS) and additional self-developed items. Higher scores indicated higher levels of self-efficacy for medication adherence.
Delivery of the intervention in everyday context | through study completion, an average of 1 year
  Quantitative assessement of intervention steps and content measured with a self-developed checklist for health care professionals
Satisfaction of HCPs with the intervention | through study completion, an average of 1 year
  Qualitative assessment (semi-structured interviews) measuring to which extend HCPs perceive the intervention as acceptable practical and sustainable
Satisfaction of patients with the intervention | through study completion, an average of 1 year
  Qualitative assessment (semi-structured interviews) measuring patient experiences with the intervention regarding acceptability and feasibility

SECONDARY OUTCOMES:
(preliminary) intervention effects on adherence | 1 year
  days of missed medication
(preliminary) intervention effects on physical activity | change from baseline at 6 and 12 months
  assessing habitual activity with the Short Questionnaire to Assess Health-enhancing physical activity (SQUASH). Higher scores indicate more time spended on habitual physical activity.
(preliminary) intervention effects on quality of life | change from baseline at 12 months
  assessed with the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES). Higher values reflect a better quality of life.
(preliminary) intervention effects on social support | change from baseline at 12 months
  assessed with the Sociale Steun Lijst - Discrepanties (SSL-D). A higher score indicates a higher lack of social support.
(preliminary) intervention effects on self-management | change from baseline at 12 months
  assessed with the Patient Activiation Measurement (PAM-13). A higher score indicates a higher level of self-management.
Treatment as usual | through study completion, an average of 1 year
  Treatment as usual will be assessed by the Treatment as usual questionnaire (an open ended questionnaire) in HCPs
Satisfaction of patients with usual care | through study completion, an average of 1 year
  qualitative semi-structured interviews with participants of the control group about their experiences of delivered care

CONTACTS AND LOCATIONS:
Locations (1):
- Bernhoven, Uden, Netherlands

IPD SHARING:
Plan to Share IPD: No